CLINICAL TRIAL: NCT03278561
Title: General Risk Factors and Inflammatory Determinants in Older Patients With Asthma
Acronym: GRANDMA
Status: Completed | Type: Observational
Sponsor: Gerdien Tramper (Other)
Responsible Party: Sponsor-Investigator, Gerdien Tramper, MD PhD, Franciscus Gasthuis
Organization: Franciscus Gasthuis (Other)
Other Study IDs: GRANDMA
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Asthma; Late-Onset Asthma; Childhood Asthma
Keywords: asthma; age of onset; inflammation; comorbidity; microbiome
MeSH Terms: conditions — Asthma; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum, blood, NP swab, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early onset asthma: Sputum induction according to the European Respiratory Society (ERS) protocol. A blood sample of 100ml will be taken.
  Interventions: Procedure: Sputum induction; Procedure: Blood sample
- Late onset asthma: Sputum induction according to the ERS protocol. A blood sample of 100ml will be taken.
  Interventions: Procedure: Sputum induction; Procedure: Blood sample
- No pulmonary disease: Sputum induction according to the ERS protocol. A blood sample of 100ml will be taken.
  Interventions: Procedure: Sputum induction; Procedure: Blood sample

INTERVENTIONS:
Procedure: Sputum induction — Sputum induction according to the ERS protocol
Procedure: Blood sample — A blood sample of 100ml will be taken.

SUMMARY:
A cross-sectional study in asthma patients to determine if a late age of onset asthma (start symptoms >18 years old), is associated with more persistent airway/systemic inflammation, worse asthma control, more co-morbidity, a different microbiome and poorer quality of life despite the use of optimized asthma therapy.

DETAILED DESCRIPTION:
For ages, asthma has been considered a disease for children and young adults. However, nowadays 30% of all asthma patients is over 50 years old. Asthma in the elderly is generally more severe and approximately 50% of all deaths drom asthma occur in this age group. With rapid aging of the global population, the burden of asthma in the elderly will further increase.

Asthma is a heterogeneous disease and the question is whether asthma in the elderly can be considered the same disease as asthma in children and young adults. The pathophysiology and risk factors of asthma in the elderly are still not completely understood. Good characterization of asthma in the elderly requires clinical phenotyping as well as a thorough analysis of the underlying cellular and molecular mechanisms. It is hypothesized that in older asthma patients, a late age of onset (start asthma symptoms >18 years) is associated with more persistent airway/systemic inflammation, worse asthma control, more co-morbidity and poorer quality of life despite the use of optimized asthma therapy.

ELIGIBILITY:
Inclusion Criteria Asthma patients:

* Age between 18-80 years
* Smoking history of < 10 packyears (PY)
* Willing and able to comply with the study protocol
* Asthma diagnosis is based on presence of typical clinical symptoms, reversible airway obstruction (+12% improvement in forced expiratory volume at one second (FEV1) after bronchodilator) or bronchial hyperreactivity (PC20 < 8 mg/ml) or a (fractional exhaled nitric oxide) FeNO > 50 ppb. - All asthma patients have (Global Initiative for Asthma ) GINA step 4-5 medication (high dose ICS/LABA).
* Asthma control questionaire (ACQ) > 0,75
* Written informed consent.

Inclusion Criteria Healthy controls:\Inclusion criteria healthy control:

* Written informed consent
* Age between 18-80 years.

Exclusion Criteria:

* Smoking history of > 10 PY
* Age < 18 years or > 80 years
* Not able to speak or write Dutch language.
* Not able to perform lung function test/sputum induction
* ACQ < 0,75
* Other diseases which could influence pulmonary function and/or the immune system such as: o A possible infection of the upper- or lower respiratory tract 4 weeks prior to the collection of materials;

  * Chronic obstructive pulmonary disorder (COPD) in the medical history;
  * Auto-immune diseases such as systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), myasthenia gravis or Goodpasture's syndrome;
  * Malignancies;
  * Inherited or acquired immunodeficiency
  * Pregnancy;

Exclusion criteria healthy controls:

* Asthma, as defined earlier (page 13);
* An abnormal spirometry with a forced vital capacity (FVC) or FEV1 below the 80% of the predicted value
* A liaison with the coordinating or principal investigator, which could likely influence the decision to participate in this study voluntarily (in concordance with the World Meteorological Organization (WMO) -article 5);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim is to enrol 30 patients with early onset asthma (age of onset < 18 years) and 30 patients with late onset asthma (age of onset > 18 years); all with a smoking history of < 10 PY. Both groups consist of 15 older asthma patients (> 50 years) and 15 younger asthma patients (< 50 years); per age group 15 healthy controls serve as comparison (no asthma). Asthma diagnosis is based on presence of typical clinical symptoms, reversible airway obstruction (+12% improvement in FEV1 after bronchodilator) or bronchial hyperreactivity (PC20 < 8 mg/ml) or a FeNO > 50 ppb. All asthma patients have GINA step 4-5 medication (high dose ICS/LABA) and are not adequately controlled (ACQ > 0,75)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in number and activation status of inflammatory cells in sputum and blood | 1 month
  To compare the differences in number and activation status of inflammatory cells in sputum and blood of different subgroups of asthmatics.)

SECONDARY OUTCOMES:
Interleukin cell type 2 (ILC2) correlation and disease phenotype | 1 month
  To find correlations between ILC2 numbers and characteristics and immunological and clinical disease phenotype. -
Hair cortisol | 1 month
  Detection of cortisol levels in hair, to determine a possible method to check Inhaled corticosteroid (ICS) adherence.
Inflammatory profile | 1 month
  To measure physiological factors (lung function, activity level) and relate them to inflammatory profile.
Selfmanagement / coping strategies | 1 month
  To investigate the relationship between duration and onset of asthma and self-management/coping strategies of patients.
The effect of aging on inflammation, physiology, psychology and co-morbidities in asthma. | 1 month
  The effect of aging on inflammation, physiology, psychology and co-morbidities in asthma.
Detection of different microbiome subgroups of asthmatics and compare with controls. | 1 month
  Detection of microflora/microbiome pattern in sputum and faeces in different subgroups of asthmatics and compare with controls.

CONTACTS AND LOCATIONS:
Overall Officials: GM de Boer, MD, Principal Investigator — Franciscus Gasthuis Rotterdam; GJ Braunstahl, MD, PhD, Principal Investigator — Franciscus Gasthuis Rotterdam; GA Tramper, MD, PhD, Principal Investigator — Franciscus Gasthuis Rotterdam
Locations (1):
- Franciscus Gasthuis, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided